CLINICAL TRIAL: NCT02700945
Title: Stroke AF - Rate of Atrial Fibrillation Through 12 Months in Patients With Recent Ischemic Stroke of Presumed Known Origin
Brief Title: Rate of Atrial Fibrillation Through 12 Months in Patients With Recent Ischemic Stroke of Presumed Known Origin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Stroke AF
Record Dates: First submitted 2016-03-02; First posted 2016-03-07 (Estimated); Results first posted 2021-11-09 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-04

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to the continuous monitoring arm or the control arm. Subjects randomized to the continuous monitoring arm will have a Reveal LINQ ICM inserted within 10 days of the qualifying stroke and undergo continuous remote monitoring. Subjects randomized to the control arm will be followed per site specific standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Reveal LINQ™ Insertable Cardiac Monitor (Active Comparator): Subjects randomized to the Reveal LINQ™ Insertable Cardiac Monitor arm will be continuously monitored via the inserted Reveal LINQ™ device.
  Interventions: Device: Reveal LINQ™ Insertable Cardiac Monitor
- Control Arm (No Intervention): Subjects randomized to the control arm will be followed per site specific standard of care.

INTERVENTIONS:
Device: Reveal LINQ™ Insertable Cardiac Monitor — The Medtronic Reveal LINQ™ ICM is a programmable device that continuously monitors a patient's ECG (electrocardiogram) and other physiological parameters. The device records cardiac information in response to automatically detected arrhythmias and patient activation.
  Other Names: LINQ; LINQ™
  Arms: Reveal LINQ™ Insertable Cardiac Monitor

SUMMARY:
The purpose of the Stroke AF study is to compare the incidence of atrial fibrillation (AF) through 12 months between continuous cardiac rhythm monitoring with the Reveal LINQ™ Insertable Cardiac Monitor (ICM) (continuous monitoring arm) and standard of care (SoC) medical treatment (control arm) in subjects with a recent ischemic stroke of presumed known origin.

DETAILED DESCRIPTION:
Stroke AF is a prospective, multi-site, randomized, controlled, non-blinded, post-market study. The Stroke AF study will compare the incidence rate of atrial fibrillation through 12 months between the continuous monitoring arm and the control arm in subjects with a recent ischemic stroke of presumed known origin. Subjects randomized to the continuous monitoring arm will have a Reveal LINQ Insertable Cardiac Monitor inserted within 10 days of the qualifying stroke and undergo continuous remote monitoring. Subjects randomized to the control arm will be followed per site specific standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had an ischemic stroke believed to be due to small vessel disease, large vessel cervical or intracranial atherosclerosis within the past 10 days
* Subject is willing and able to undergo study requirements and expected to be geographically stable during study follow-up
* Subject is 60 years of age or older, or age 50 to 59 years plus a documented medical history of at least one of the following additional risk factors for stroke:

  * Congestive heart failure
  * Hypertension (Systolic Blood Pressure > 140)
  * Diabetes Mellitus
  * Prior Stroke (>90 days ago, other than study qualifying index event)
  * Vascular disease (e.g. coronary artery disease, heart attack, peripheral artery disease and complex aortic plaque)

Exclusion Criteria:

* Subject has had a cryptogenic stroke
* Subject has had a cardioembolic stroke
* Subject has untreated hyperthyroidism
* Subject has had a recent myocardial infarction <1 month of stroke
* Subject has had a recent cardiac surgery (e.g. coronary artery bypass surgery (CABG)) <1 month of stroke
* Subject has a mechanical heart valve
* Subject has valvular disease requiring immediate surgical intervention
* Subject has documented prior history of atrial fibrillation or atrial flutter
* Subject has permanent indication for oral anticoagulation
* Subject has permanent contraindication to oral anticoagulation such that detection of AF would not change medical management, based on enrolling investigators judgment
* Subject is enrolled in a concurrent study that may confound the results of this study. Co-enrollment in any concurrent clinical study (including registries) requires approval of the study manager or designee.
* Subject's life expectancy is less than 1 year
* Subject is pregnant
* Subject has or is indicated for implant with a pacemaker, Implantable Cardioverter Defibrillator (ICD), Cardiac ResynchronizationTherapy (CRT), or an implantable hemodynamic monitor
* Subject with a medical condition that precludes the patient from participation in the opinion of the investigator

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bernstein, PhD/MD, Study Chair — Northwestern University; Lee Schwamm, MD, Study Chair — Mass General
Locations (35):
- United States (35):
  - Cardiovascular Associates of the Southeast, Birmingham, Alabama
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - University of California San Francisco UCSF Medical Center, San Francisco, California
  - Innovative Medical Research of South Florida, Aventura, Florida
  - University of Miami Hospital, Miami, Florida
  - AdventHealth Neuroscience Institute, Orlando, Florida
  - The Queens Medical Center, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Neuroscience Institute, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Health Partners Institute (Bloomington MN), Bloomington, Minnesota
  - Health Partners Institute (Saint Louis Park MN), Saint Louis Park, Minnesota
  - Cox Medical Center South, Springfield, Missouri
  - Mercy Clinic Cardiology, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Albany Medical Center, Albany, New York
  - University at Buffalo, The State University of New York, Buffalo, New York
  - North Shore University Hospital, New Hyde Park, New York
  - NYU Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Overlook Medical Center, Summit, New York
  - Cone Health, Greensboro, North Carolina
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - PeaceHealth Sacred Heart Medical Center at Riverbend, Springfield, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - Saint Thomas Research Institute, Nashville, Tennessee
  - Baylor Research Institute Dallas - Baylor University Medical Center (BUMC), Dallas, Texas
  - University of Texas (UT) Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Centra Medical Group Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
This data is for internal, Medtronic use only. Data from the study will be analyzed and submitted in the form of abstracts and possible publication in a journal.

REFERENCES:
- [Derived] Bernstein RA, Kamel H, Granger CB, Piccini JP, Katz JM, Sethi PP, Pouliot E, Franco N, Ziegler PD, Schwamm LH; STROKE AF Investigators. Atrial Fibrillation In Patients With Stroke Attributed to Large- or Small-Vessel Disease: 3-Year Results From the STROKE AF Randomized Clinical Trial. JAMA Neurol. 2023 Dec 1;80(12):1277-1283. doi: 10.1001/jamaneurol.2023.3931. PMID 37902733
- [Derived] Schwamm LH, Kamel H, Granger CB, Piccini JP, Katz JM, Sethi PP, Sidorov EV, Kasner SE, Silverman SB, Merriam TT, Franco N, Ziegler PD, Bernstein RA; STROKE AF Investigators. Predictors of Atrial Fibrillation in Patients With Stroke Attributed to Large- or Small-Vessel Disease: A Prespecified Secondary Analysis of the STROKE AF Randomized Clinical Trial. JAMA Neurol. 2023 Jan 1;80(1):99-103. doi: 10.1001/jamaneurol.2022.4038. PMID 36374508
- [Derived] Zachrison KS, Amati V, Schwamm LH, Yan Z, Nielsen V, Christie A, Reeves MJ, Sauser JP, Lomi A, Onnela JP. Influence of Hospital Characteristics on Hospital Transfer Destinations for Patients With Stroke. Circ Cardiovasc Qual Outcomes. 2022 May;15(5):e008269. doi: 10.1161/CIRCOUTCOMES.121.008269. Epub 2022 Apr 4. PMID 35369714
- [Derived] Bernstein RA, Kamel H, Granger CB, Piccini JP, Sethi PP, Katz JM, Vives CA, Ziegler PD, Franco NC, Schwamm LH; STROKE-AF Investigators. Effect of Long-term Continuous Cardiac Monitoring vs Usual Care on Detection of Atrial Fibrillation in Patients With Stroke Attributed to Large- or Small-Vessel Disease: The STROKE-AF Randomized Clinical Trial. JAMA. 2021 Jun 1;325(21):2169-2177. doi: 10.1001/jama.2021.6470. PMID 34061145

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We enrolled 496 participants in the study but only 492 were randomized. Three participants were enrolled but did not meet eligibility criteria, the fourth withdrew consent.
Period: Overall Study
Arm/Group | Reveal LINQ™ Insertable Cardiac Monitor | Control Arm
Started | 242 | 250
Completed | 210 | 207
Not Completed | 32 | 43

BASELINE CHARACTERISTICS:
Population: Two participants in the 'continuous monitoring' arm of the study did not collect baseline information after randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Reveal LINQ™ Insertable Cardiac Monitor | Control Arm | Total
Number analyzed (Participants) | 240 | 250 | 490
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 117 | 113 | 230
  >=65 years | 123 | 137 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (9.3) | 67.5 (9.5) | 67.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 89 | 185
  Male | 144 | 161 | 305
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 240 | 250 | 490
Tobacco Use [Count of Participants; unit: Participants] | 130 | 133 | 263
Congestive Heart Failure [Count of Participants; unit: Participants] | 28 | 23 | 51
Hypertension [Count of Participants; unit: Participants] | 197 | 200 | 397
Stroke/TIA/Thromboembolism [Count of Participants; unit: Participants] | 240 | 250 | 490
Vascular Disease [Count of Participants; unit: Participants] | 45 | 47 | 92

OUTCOME MEASURES:

1. Primary Outcome: The Rate of AF Through 12 Months in Subjects With a Recent Ischemic Stroke of Presumed Known Origin.
Description: AF will be defined as an AF event lasting more than 30 seconds. The first AF episode detected and adjudicated by the endpoint adjudication committee will be used for this analysis.
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Reveal LINQ™ Insertable Cardiac Monitor | Control Arm
Number analyzed (Participants) | 242 | 250
percentage of participants | 12.5 | 1.8
Statistical Analysis 1: Comparison: Reveal LINQ™ Insertable Cardiac Monitor vs Control Arm; H0: h(t) = hT(t) for t ≤ 12 months HA: hC(t) ≠ hT(t) for t ≤ 12 months where hT(t) and hC(t) are the hazard functions of first detected and adjudicated AF at time t for subjects with and without the Reveal LINQ diagnostics for AF, respectively. Hazard functions and survival functions are transformations of each other; Test type: Superiority — The 12-month Kaplan-Meier estimate will be reported for each arm. The hazard ratio estimate for the treatment effect with its 95% confidence interval will be reported; p < 0.001, Log Rank — A priori threshold is .05; Hazard Ratio (HR) = 7.4, 95% CI 2-sided [2.6 to 21.3] — A hazard ratio of > 1 indicates that continuous monitoring arm is superior to control arm in detecting AF

2. Secondary Outcome: The Rate of AF Through the Duration of Study Follow-up (36 Months) Between Study Arms.
Description: as for outcome 1
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Reveal LINQ™ Insertable Cardiac Monitor | Control Arm
Number analyzed (Participants) | 242 | 250
percentage of participants | 21.7 | 2.4

ADVERSE EVENTS:
Time Frame: We monitored adverse events up to the primary end point from enrollment, which was equivalent to 1 year.
Arm/Group | Reveal LINQ™ Insertable Cardiac Monitor | Control Arm
All-Cause Mortality (participants affected / at risk) | 5/242 | 12/250
Serious Adverse Events (participants affected / at risk) | 58/242 | 65/250
Other Adverse Events (participants affected / at risk) | 69/242 | 45/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reveal LINQ™ Insertable Cardiac Monitor (N=242) | Control Arm (N=250)
Accelerated hypertension (Vascular disorders) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 7 (9) | 6 (7)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 7 (7)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Basal ganglia stroke (Nervous system disorders) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 3 (4)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac stress test abnormal (Investigations) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 10 (10) | 12 (12)
Cerebral infarction (Nervous system disorders) | 1 (1) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 5 (5)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3) | 6 (6)
Death (General disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 2 (3) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Hypertensive urgency (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 2 (2)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 11 (13) | 14 (14)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Lupus endocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Stroke in evolution (Nervous system disorders) | 1 (1) | 1 (1)
Subclavian steal syndrome (Vascular disorders) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 2 (2)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 3 (4)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Vertebral artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reveal LINQ™ Insertable Cardiac Monitor (N=242) | Control Arm (N=250)
Angina pectoris (Cardiac disorders) | 2 (2) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 30 (30) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 4 (4) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
C-reactive protein abnormal (Investigations) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 13 (13) | 18 (19)
Hypotension (Vascular disorders) | 1 (1) | 6 (6)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Implant site pain (General disorders) | 1 (1) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 3 (3) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Stroke in evolution (Nervous system disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 4 (4)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 2 (2)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The attribution of stroke mechanism is subjective and may have led to the enrollment of a population at higher risk of underlying embolism. However, this attribution reflects real-world practice and our sample is representative of patients in whom ICM decisions need to be made. The assignment to ICM versus control was not blinded, however our study endpoint was adjudicated using objective criteria. Our study was not powered to detect a significant difference in rates of recurrent stroke.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT02700945/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT02700945/SAP_001.pdf